CLINICAL TRIAL: NCT04865315
Title: HiLoGlio Organoid Study: 'A Living Tissue Bank of Patient-Derived Organoids From Glioma Tumors'
Brief Title: A Living Tissue Bank of Patient-Derived Organoids From Glioma Tumors
Acronym: HiLoGlio
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); Zuyderland Medisch Centrum (Other); Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Other Study IDs: HiLoGlio Organoid Study
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Low-grade Glioma; High Grade Glioma
Keywords: Prospective study; Patient-derived organoids
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low grade glioma patients: Patients who have a MRI lesion suspected for a low grade glioma (newly diagnosed or recurrent), who are eligible for a resection of the tumor
- High grade glioma patients: Patients who have a MRI lesion suspected for a high grade glioma (newly diagnosed or recurrent), who are eligible for a resection of the tumor

SUMMARY:
There is a high medical need to improve treatment outcome for high-grade and low-grade glioma since no curative treatment is available. To achieve this goal, a broader understanding is needed of the causes of inter-and intratumoral heterogeneity; glioma dedifferentiation and invasion; the major determinants of malignancy and treatment failure in glioma patients. Patient-derived organoid (PDOs) of high-grade gliomas and low-grade gliomas will be used to identify the mechanisms that underlie this malignant behaviour and treatment resistance. This insight may be used to develop patient avatars to simultaneously test multiple new treatment modalities that are predictive for survival and quality of life of glioma patients.

DETAILED DESCRIPTION:
To establish primary patient-derived three-dimensional organoid cultures from low grade and high-grade gliomas to study the mechanisms that contribute to i.e.

resistance to radiotherapy and/or chemotherapy and immunotherapy, dedifferentiation, tumor invasion among others, in primary and recurrent tumors.

Primary Objectives:

1. Establishment of primary patient-derived organoids (PDO) of 'de novo' and recurrent high-grade glioma (HGG) and low-grade glioma (LGG)
2. Phenotypic, genetic, epigenetic and transcriptomic characterization of HGG and LGG organoids and resemblance to the parental tumor (i.e. characterization of specific cell populations and genomic and transcriptomic profiles of PDOs)
3. Investigation of combinations of new or standard glioma systemic treatments (i.e immunotherapy, chemotherapy) with or without radiation (i.e. protons, photons).

Secondary objectives

1. Establishment of co-cultures of HGG and LGG organoids with immune cells.
2. Investigation of radiation-triggered cell death mechanisms on PDOs after irradiation with photons and protons.
3. Investigation of dedifferentiation mechanisms of LGG to HGG in the context of radiation w/wo immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* MRI diagnosis of low grade glioma (LGG) or high grade glioma (HGG)
* Age 18 years or older
* Patient is eligible for a resection of the tumor

Exclusion Criteria:

* Contra-inidication for neurosurgical resection of the tumor.
* Incapacitated patient, unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have an MRI lesion suspected for a low- or high grade glioma (newly diagnosed or recurrent), who are eligible for a resection of the tumor.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Phenotypic, genetic, epigenetic proteomic and transcriptomic profile of the LGG/HGG PDOs | Baseline tumor resection and blood sampling
  Phenotypic, genetic, epigenetic proteomic and transcriptomic profile of the LGG/HGG PDOs will be performed after establishing PDO and the data will be compared with the phenotypic, genetic, epigenetic, proteomic and transcriptomic profile of the parental tumor. DNA isolated from peripheral blood will be used as normal reference DNA for (epi)genetic profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vooijs, Prof. Dr., Principal Investigator — Maastro Radiaton Oncology clinic
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
All obtained research data points and information will be added in a coded manner to the existing database of Laboratory Radiotherapy, located on a MUMC+ hosted and secured server and is password protected. A dedicated, trained person will add all genetic and research information from this project to the database, which was especially designed for this research. Only coded information will be extracted and used for the downstream research analyses.